CLINICAL TRIAL: NCT01200043
Title: Metabolic Impact of Fructose Restriction in Obese Children
Acronym: SUCRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Touro University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSF-2845; R01DK089216 (NIH)
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Obesity; Metabolic Syndrome
Keywords: Childhood obesity; metabolic syndrome; insulin resistance; intrahepatic fat; hypertension
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Pediatric Obesity; Insulin Resistance; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- fructose restriction (Experimental): Isocaloric fructose restricted diet for 10 days
  Interventions: Other: fructose restriction diet

INTERVENTIONS:
Other: fructose restriction diet — fruits and vegetables only

SUMMARY:
The sugar fructose has been implicated not just as a cause of obesity, but as a cause of the metabolic diseases that go along with obesity, termed "metabolic syndrome". Obese children with metabolic disease will be studied before and after 10 days of a fructose restricted diet. The question is whether their co-morbidities will improve, even if weight remains constant.

DETAILED DESCRIPTION:
Recent studies suggest that specific types of macronutrients in the diet may have selective effects on nutrient absorption, insulin sensitivity, and lipid metabolism. Elucidation of the metabolic impact of specific dietary components may well result in improved efficacy of lifestyle approaches to reduce obesity and metabolic diseases. Despite similar fructose consumption, the phenotype of co-morbidities is different between African Americans and Latinos. Latino and Caucasian children manifest worsened dyslipidemia and non-alcoholic fatty liver disease (NAFLD), while African American children manifest worsened insulin resistance and hypertension. We have also documented in adults that a reduction in de novo lipogenesis (DNL; production of new lipids) in the liver and liver fat content, and improvement in hepatic insulin sensitivity were achieved by substitution of complex carbohydrate for fructose; but these changes appeared less dramatic in African American compared to Latino or Caucasian subjects. These divergent findings suggest ethnic and race-specific differences of fructose metabolism and disposition.

To determine whether fructose is a contributor to metabolic co-morbidity in children, we will conduct a convenience cohort within-subject intervention with repeated measures, stratified by racial/ethnic group (Latinos vs. African Americans vs. Caucasians). The intervention will consist of restricting fructose ingestion only to naturally-occurring fructose in fruits and vegetables (approximately 15 gm/day for 10 days), by substituting complex carbohydrate for excess dietary fructose, while maintaining neutral energy balance. We anticipate fructose restriction to differentially improve co-morbidities in different racial/ethnic groups.

ELIGIBILITY:
Inclusion Criteria:

* African-American, Latino, and Caucasian boys and girls. Ethnicity is to be determined by self-report. Utilizing the US Census Bureau procedures, participants will be asked two questions, the first regarding ethnicity and the second on race. Subjects will be given the opportunity to select more than one racial category.
* Ages 8 to 18 yr. The minimum age cutoff is due to our desire not to sedate younger children for the magnetic resonance spectroscopy scan or magnetic resonance scan (MRS, MRI). We chose to study these groups because they are most affected by metabolic syndrome and manifest the greatest morbidities; yet their presentations are different from each other.
* The following criteria are modified from the National Cholesterol Education Program's Adult Treatment Panel and the World Health Organization definition of metabolic syndrome. Waist circumference is not an adequate predictor of visceral adiposity in children. Also, no normative values have been developed nor is this measurement consistent between racial and ethnic groups. Body mass index (BMI), however, correlates strongly with both visceral lipid depot and blood pressure. The definition of hypertension is greater than the 95th percentile for sex and age as designated in the 1996 Task Force Report on High Blood Pressure in Children and Adolescents.

  1. Obesity, as defined by BMI z-score of 2.0 or greater, or above the 97th percentile for age and sex; and weight ≥40 kg.
  2. Hyperinsulinemia (fasting insulin >15 µU/mL), or insulin resistant (HOMA > 4.3). See details below.
  3. At least one of the following: systolic blood pressure above the 95th percentile for age and sex, or triglyceride level above the 95th percentile for age, sex and race or ethnic group as established by the 1998 National Heart, Lung, and Blood Institute Growth and Health Study.

Exclusion Criteria:

* History of disorders other than obesity that may affect insulin levels, such as Cushing's syndrome, diabetes mellitus, or depression.
* Medications that may affect insulin sensitivity or hepatic lipid content, e.g. metformin, steroids, atypical antipsychotics, anti depressants, statins, Vitamin E, thyroid medications, anti-hypertensives, weight loss medications, oral contraceptives.
* Pregnancy or lactation.
* Surgical procedures for obesity.
* History consistent with obstructive sleep apnea.
* Implants including intracranial surgical clips, pacemakers, and other metals or implants that preclude MR scanning.
* Claustrophobia.
* Inability to fit within the MR bore: shoulder to shoulder width of greater than 58 cm or anterior-posterior length greater than 35 cm (magnet bore size limitation).
* Weight greater than 320 pounds (MRS table weight limitation).
* Eating disorders.
* Smoking or alcohol use. Subjects will answer the two questions on the Alcohol Query Form. Any consumption of more than 2 drinks per month will
* Vegan diet.
* All subjects with known diabetes mellitus according to the 1997 ADA criteria will be excluded. However, subjects with known impaired glucose tolerance (fasting glucose 101-125, and 2-hour post-prandial glucose level between 141-200) can remain eligible.
* Syndromic patients (e.g. Prader-Willi, Bardet-Biedl) will be excluded, as it is likely that the reasons for their obesity may be neurologic or single-point mutations, and are likely to be different from those causing the Metabolic Syndrome.
* Subjects who are found to be hypothyroid by clinical exam or by evaluation of thyroid function tests on first visit to the WATCH Clinic will receive L-thyroxine for three months, with documentation of adequate replacement, prior to enrollment in the protocol.
* Subjects with a history of hepatitis will be excluded from the study. However, patients with NAFLD, as determined by Dr. P. Rosenthal (Ped. Hepatology, UCSF), may participate. Upper cutoffs for AST and ALT will be 5 times the upper limit of normal for the UCSF laboratory.
* Subjects with any history of renal disease will be excluded.
* Subjects who have a fever or an active infection will be postponed until their infection remits.
* Emancipated minors will be excluded, as there will be no parental supervision and monitoring over the subject's diet during the 9 days of fructose restriction.
* Females who have achieved menarche will have a urine pregnancy test at the time of their DEXA scans. A positive pregnancy test will lead to exclusion of the data from further analysis. Results of a positive pregnancy test will be transmitted to the minor only, and the parents will be told only that the subject does not qualify for the study.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2010-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12-01 (Actual)

PRIMARY OUTCOMES:
intrahepatic fat content | 10 days
  We anticipate fructose restriction to reduce intrahepatic fat, exclusive of calories

SECONDARY OUTCOMES:
insulin resistance | 10 days
  We anticipate fructose restriction will improve insulin sensitvity exclusive of calories

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lustig, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

REFERENCES:
- [Derived] Schwarz JM, Noworolski SM, Erkin-Cakmak A, Korn NJ, Wen MJ, Tai VW, Jones GM, Palii SP, Velasco-Alin M, Pan K, Patterson BW, Gugliucci A, Lustig RH, Mulligan K. Effects of Dietary Fructose Restriction on Liver Fat, De Novo Lipogenesis, and Insulin Kinetics in Children With Obesity. Gastroenterology. 2017 Sep;153(3):743-752. doi: 10.1053/j.gastro.2017.05.043. Epub 2017 Jun 1. PMID 28579536
- [Derived] Gugliucci A, Lustig RH, Caccavello R, Erkin-Cakmak A, Noworolski SM, Tai VW, Wen MJ, Mulligan K, Schwarz JM. Short-term isocaloric fructose restriction lowers apoC-III levels and yields less atherogenic lipoprotein profiles in children with obesity and metabolic syndrome. Atherosclerosis. 2016 Oct;253:171-177. doi: 10.1016/j.atherosclerosis.2016.06.048. Epub 2016 Jul 19. PMID 27451002